CLINICAL TRIAL: NCT03668743
Title: Pregnancy Loss Between 15 and 22 Weeks SA Within the Network of Perinatal Period of Western Brittany : Case Control Study
Brief Title: Pregnancy Loss Between 15 and 22 Weeks SA Within the Network of Perinatal Pérriodof Western Brittany : Case Control Study PILOT STUDY CA
Acronym: PEGREP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PEGREP (29BRC17.0056)
Record Dates: First submitted 2018-09-11; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2017-05

CONDITIONS: Miscarriage in Second Trimester
Keywords: risk factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The etiologies and some risk factors for pregnancy loss in the 2nd trimester are described in the literature. However, there are some risk factors that are not studied. The PEGREP study is a retrospective observational case-control study whose main objective is to identify risk factors for pregnancy loss between 15 and 22 weeks. The patients included cases are women who had a pregnancy loss between 15 and 22 SA between 2010 and 2015 and who were listed during the mortality reviews of the perinatal network of Western Brittany. The patient witnesses gave birth at the end of a healthy child in one of the maternity of Western Brittany. Matching 1 case for 1 controls was done on the woman's age, parity and number of fetuses.

DETAILED DESCRIPTION:
The etiologies of late miscarriages are well described in the literature. Globally, these are premature deliveries, namely: malformations of the genital tract (uterine malformations, cervico-isthmic incompetence), infections (chorioamniotitis, cervico-vaginal infections) and fetal causes (hydramnios, multiple pregnancies). Some risk factors are also described as extreme maternal age (<16 years,> 35 years), social deprivation, sleep deprivation, smoking, prenatal diagnosis, Fake's antecedent Delayed diapers (FCT), premature rupture of membranes, premature delivery or conization.

The etiologies of Fetal Deaths In Utero (MFIU) are also described: placental abnormalities, funicular abnormalities, fetal-maternal haemorrhage, fetal abnormalities (malformations, aneuploidy, genetic abnormalities), infections (in particular strepto B, E. coli and toxoplasmosis).

Certain risk factors are not studied in terms of their influence on fetal loss: body mass index (BMI), existence of chronic pathologies (diabetes, thyroid diseases, depression, other chronic diseases, etc.). ..), uterine scarring, uterine endoscopic surgery ATCD, sterility treatment (induction of ovulation, procreation medical assistance (MPA) type insemination or IVF, 1st trimester bleeding, prenatal diagnosis procedure (amniocentesis or biopsy trophoblast).

population concerned: Patients who had a pregnancy loss between 15 and 22 SA between 2010 and 2015, listed thanks to the data sheets of the Western Brittany Perinatal Network

Main objective: To identify risk factors for pregnancy loss between 15 SA and 22 SA.

main endpoint: BMI, existence of chronic pathologies (diabetes, thyroid pathologies, depression, other chronic diseases .....), treatments, uterine scarring, antecedent of uterine endoscopic surgery, treatment of infertility (induction of ovulation, medical assistance in procreation (MPA) type insemination or IVF), first trimester bleeding, prenatal diagnosis procedure (amniocentesis or trophoblast biopsy).

Methodology: Retrospective multicenter case-control study. Pairing 1 case for 1 witnesses. Match with age, parity, number of fetuses (single or multiple pregnancy)

Statistics: A typical descriptive analysis will be performed (means and standard deviation, medians and quartiles, proportions). Comparisons will be performed univarially by a matched Chi-square for proportions, a paired Student T-test if normal distribution or a matched non-parametric test (matched Willcoxon test) if non-normal distribution. Then a multivariate analysis will be performed using conditional logistic regression.

Criteria for inclusion:

CAS:

* patients who had a pregnancy loss between 15 and 22 SA between 2010 and 2015
* having given birth in one of the maternities of Western Brittany
* listed during the mortality reviews of the perinatal network of Western Brittany.

WITNESSES:

* patients who have given birth (> 37SA) of healthy children
* having given birth in one of the maternity of Western Brittany. Pairing: Age, parity, number of fetuses (single or multiple pregnancy). Pairing 1 case for 1 witnesses.

Listed at Brest CHRU

Exclusion criteria:

* Pregnancy loss after 22 weeks,
* medical or therapeutic interruptions of pregnancy, fetuses whose anatomopathology describes biometrics below 15SA, fetuses with chromosomal malformations or abnormalities diagnosed before pregnancy loss.

Number of patients: 101 cases, 101 controls. The number of cases identified is 101, and the number of controls is set at 101 (1: 1).

Expected benefits: This study will identify or suggest high-intensity risk factors (OR> 4); but the study will not be powerful enough to identify possible factors of lesser intensity (OR <2). These preliminary results will lead to the subsequent development of a prospective study adjusted to specific and quantified hypotheses in order to establish an adequate number of necessary subjects.

ELIGIBILITY:
Inclusion Criteria:

CAS:

* patients who had a pregnancy loss between 15 and 22 SA between 2010 and 2015
* having given birth in one of the maternities of Western Brittany
* listed during the mortality reviews of the perinatal network of Western Brittany.

WITNESSES:

* patients who have given birth (> 37SA) of healthy children
* having given birth in one of the maternity of Western Brittany. Pairing: Age, parity, number of fetuses (single or multiple pregnancy). Pairing 1 case for 1 witnesses.

Listed at Brest CHRU

Exclusion Criteria:

* Pregnancy loss after 22 weeks,
* medical or therapeutic interruptions of pregnancy,
* fetuses whose anatomopathology describes biometrics below 15SA,
* fetuses with chromosomal malformations or abnormalities diagnosed before pregnancy loss.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had a loss of pregnancy between 15 and 22 SA between 2010 and 2015, listed thanks to the data sheets of the perinatal network of Western Brittany
Sampling Method: Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
maternal history | at the time of diagnosis of fetal loss (Day1)
  chronic diseases, history of gynecology and obstetrics
criteria of the pregnancy concerned by the fetal loss | at the time of diagnosis of fetal loss ( Day 1)
  pregnancy after infertility treatment, antenatal invasiveness, 1st trimester, premature bleeding, gestational diabètes, rupture of membranes

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure SALAUN, Principal Investigator — University Hospital, Brest
Locations (2):
- France (2):
  - SALAUN Anne -Laure, Brest
  - CHRU de Brest, Brest